CLINICAL TRIAL: NCT01298375
Title: Metabolic Characterization of Type 2 Diabetic, Obese, Lean Sedentary and Endurance Trained Individuals in Vivo, ex Vivo and in Vitro
Brief Title: Metabolic Phenotyping in Humans
Acronym: MetPhe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL35178.068.11
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Healthy; Obesity; Type 2 Diabetes Mellitus
Keywords: Metabolic flexibility; Mitochondrial function; Human primary myoblasts; Lipid metabolism
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, RNA, tissue, primary myoblasts, mitochondria
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Type 2 diabetes (T2D) is a global burden disease affecting almost 200 million people and is expected to nearly double by 2030 (1). It is imperative that this disease is kept under control, and that we begin to reverse the direction of its incidence. We propose to start by identifying the physiological and molecular aspects of the problem in all spectrums of the disease (ie from insulin sensitive athletes to sedentary lean and obese individuals and further to overt type 2 diabetics), and focus our efforts on examining the differences and identifying the stages of progression for possible targets of future intervention. The proposed study "Metabolic Phenotyping" is novel in its target populations and innovative in its use of state-of-the-art techniques. We hypothesize that the in vivo differences in metabolic flexibility and mitochondrial function between endurance athletes and type 2 diabetics and their lean and obese controls are retained in vitro and will offer a new model in which to study the underlying mechanisms of the progression of T2D.

DETAILED DESCRIPTION:
The aim of the present research proposal is to metabolically phenotype endurance trained athletes, lean and obese sedentary and type 2 diabetic individuals with the following objectives:

1. assess metabolic flexibility as measured by a euglycemic-hyperinsulinemic clamp
2. measure in vivo mitochondrial function by MRS of phosphocreatine (PCr) recovery
3. establish primary myoblast cell lines to correlate with the above in vivo measurements, as well as further explore dietary, pharmacological and genetic manipulations in vitro
4. quantify intramyocellular lipid (IMCL) and acetylcarnitine in vivo by MRS

Study population:

A total of 132 male participants (18-70 years) will participate in this study. The first group of 33 participants will be lean endurance-trained athletes, the second group will be lean sedentary control participants, the third group will be sedentary type 2 diabetic participants, and the last group of 33 participants will be obese, non-diabetic sedentary control participants. It is preferred to use male participants in order to minimize variation in the measurements by avoiding confounding factors such as hormones.

Main study parameters/endpoints: The main study parameters are differences in metabolic flexibility as measured by euglycemic-hyperinsulinemic clamp, PCr recovery, IMCL and acetylcarnitines as measured by MRS and establishment of primary myoblast cell lines for future use.

ELIGIBILITY:
General Inclusion criteria:

* Male sex
* Generally healthy with specifically no known cardiovascular disease or gastric ulcers, which can affect the study parameters
* Stable dietary habits (no weight loss/gain > 3 kg in the last 6 months)

Group 1, type 2 diabetes participants:

* Ages 40-70 years
* BMI > 30 kg/m2
* Non-insulin dependent type 2 diabetes
* Must be on sulphonylurea (SU)-derivate or metformin therapy for at least six months with a constant dose for at least two months, or on dietary treatment for at least six months
* Well-controlled diabetes: HbA1c < 8%
* No diabetes related co-morbidities like cardiovascular diseases, diabetic foot, polyneuropathy, retinopathy

Group 2, obese healthy control participants:

* Ages 40-70 years
* BMI > 30 kg/m2
* A plasma glucose level lower than 6.1 mmol/L
* No family history of diabetes
* No medication use
* Sedentary lifestyle; No participation in any physical activity for at least 2 years

Group 3, endurance trained athletes:

* Ages 18-35 years
* BMI < 25 kg/m2
* No family history of diabetes
* No medication use
* VO2max > 55ml/kg/min
* Active in competitive endurance-exercise activities, 3 times a week for at least 2 years
* Stable level of training for at least 6 months

Group 4, lean healthy sedentary control participants:

* Ages 18-35 years
* BMI < 25 kg/m2
* No family history of diabetes
* No medication use
* VO2max < 55ml/kg/min
* Plasma glucose < 6.1 mmol/L
* Sedentary lifestyle; No participation in physical activity for more than 1 hour per week for at least 2 years

General Exclusion criteria:

* Regular smokers
* Participation in other studies
* Female sex
* Insulin dependent diabetic individuals
* Participants with diabetes related diseases (diabetic foot, diabetic polyneuropathy, diabetic retinopathy etc.)
* Use of Thiazolidines (glitazone/rosiglitazone/pioglitazone/troglitazone)
* Use of anti-coagulants (not thrombocyte-aggregation inhibitors)
* Aberrant ECG (with signs of ischemia or cardiac failure or arrythmias)
* Weight gain/loss > 3 kg in the last 6 months
* HbA1c < 7.8 in type 2 diabetic individuals
* Contraindications for MRS scans:

  * Electronic implants such as pacemakers or neurostimulator
  * Iron-containing foreign bodies in eyes or brain
  * Some hearing aids and artificial (heart) valves which are contraindicated for MRS
  * Claustrophobia
* Participants, who do not want to be informed about unexpected medical findings, or do not wish that their physician be informed, cannot participate in the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Human volunteers from the surrounding area
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2011-03; Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Euglycemic-hyperinsulinemic clamp for measurement of insulin sensitivity and metabolic flexibility | 10 hours
  After taking fasting blood samples, a primed constant infusion of glucose is initiated. Plasma glucose levels are clamped at ~5 mmol/L by variable co-infusion of 20% glucose. Every 5 minutes, blood is sampled for immediate determination of plasma glucose concentration. Glucose infusion rate is adjusted to obtain plasma glucose levels of ~5 mmol/L (euglycemia). A bolus of insulin is then infused. Before and during steady state, substrate oxidation is measured using an indirect calorimeter, which determines metabolic flexibility.

SECONDARY OUTCOMES:
Evaluating mitochondrial function through measurement of phosphocreatine (PCr) recovery by phosphorus magnetic resonance spectroscopy (31P-MRS) within the skeletal muscle | 1.5 hours
  The quantification of energy metabolites (Pi, PCr and ATP) in skeletal muscle will be performed in the v. lateralis at rest, during submaximal knee-extension exercise and during recovery. The rate at which PCr concentration is restored after exercise is an excellent in vivo measure of skeletal muscle mitochondrial oxidative capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Study Director — Maastricht University; Lauren M Sparks, PhD, Principal Investigator — Maastricht University; Madeleen Bosma, M.S., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Mancilla RF, Lindeboom L, Grevendonk L, Hoeks J, Koves TR, Muoio DM, Schrauwen P, Schrauwen-Hinderling V, Hesselink MK. Skeletal muscle mitochondrial inertia is associated with carnitine acetyltransferase activity and physical function in humans. JCI Insight. 2023 Jan 10;8(1):e163855. doi: 10.1172/jci.insight.163855. PMID 36413408
- [Derived] Houzelle A, Jorgensen JA, Schaart G, Daemen S, van Polanen N, Fealy CE, Hesselink MKC, Schrauwen P, Hoeks J. Human skeletal muscle mitochondrial dynamics in relation to oxidative capacity and insulin sensitivity. Diabetologia. 2021 Feb;64(2):424-436. doi: 10.1007/s00125-020-05335-w. Epub 2020 Nov 30. PMID 33258025